CLINICAL TRIAL: NCT01137552
Title: A Phase 1, First-in-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 780 in Adult Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Dose Escalation Study of AMG 780 in Adult Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part A, the dose escalation and primary objective of the study, was completed. Part B, the dose expansion, was not conducted due to a business decision.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070879
Record Dates: First submitted 2010-04-22; First posted 2010-06-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Advanced Solid Tumors
Keywords: First-In-Human; Dose Escalation; Dose Expansion; Advance Solid Tumors; Anti-Angiopoietin; Advance Malignancy; Cancer; Oncology; Oncology Patients; Phase 1; Clinical Trial; Tumors; Solid Tumors; Angiogenesis Inhibitors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Dose Escalation
  Interventions: Drug: AMG 780
- B (Experimental): Dose Expansion
  Interventions: Drug: AMG 780

INTERVENTIONS:
Drug: AMG 780 — AMG 780 will be administered by IV infusion every 2 weeks

SUMMARY:
This is a first in human, open-label, sequential dose escalation and expansion study of AMG 780 in up to 62 subjects with advanced solid tumors. The dose escalation part of the study is aimed at evaluating the safety, tolerability, pharmacokinetics and pharmacodynamics of AMG 780. The dose expansion will consist of up to 20 subjects and the dose level of AMG 780 will be dependent upon emerging safety and PK data from the dose escalation part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old
* Must have a pathologically documented, and definitely diagnosed, advanced solid tumor that is refractory to standard treatment, or for which no curative therapy is available, or for subjects who refuse standard therapy
* Measurable disease by RECIST criteria
* Must be able to undergo MRI evaluation
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Competent to sign and date an Institutional Review Board approved informed consent form

Exclusion Criteria:

* Presence of untreated or symptomatic primary central nervous system tumors or metastases
* Presence of leukemia or myelodysplastic syndrome
* Subjects with head and neck cancer
* Previous hematopoietic stem cell transplant (allogeneic)
* Unresolved hematological toxicities > grade 1 with the exception of grade 2 lymphopenia and non-hematological toxicities > grade 1, excluding alopecia and grade 2 neuropathy, from prior anti-cancer therapy
* Myocardial infarction within 1 year before study day 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function
* History of stroke, arterial or venous thrombosis, or pulmonary embolism within 1 year before study
* Active peripheral vascular disease
* History of bleeding diathesis
* History of pulmonary hemorrhage or gross hemoptysis within 6 months before study
* Known history of adrenal hemorrhage
* Known positive test for human immunodeficiency virus infection, or active hepatitis B or hepatitis C
* Major surgery within 1 month before study
* Prior treatment with any agent targeting the angiopoietin-Tie2 signaling pathway
* Concurrent antitumor treatment, except Lupron for subjects with prostate cancer and selective estrogen receptor modulators (SERMS) for subjects with breast cancer, within 4 weeks (6 weeks for nitrosoureas or mitomycin) before study day 1
* Known sensitivity to mammalian-derived products, bacterially-produced proteins, or any of the products to be administered during dosing
* Investigational agent within 30 days before study
* Pregnant (eg, positive urine test) or breastfeeding
* Subjects of childbearing potential, or subject who has a partner of childbearing potential, and is not using highly effective contraceptive precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AMG 780 in subjects with advanced solid malignancies (including adverse event rate, incidence of dose-limiting toxicities, and determination of maximum tolerated dose) | 2.5 years
To evaluate the pharmacokinetic (PK) parameters of AMG 780 including, but not limited to Cmax, AUC, and accumulation ratio | 2.5 years

SECONDARY OUTCOMES:
To evaluate tumor response using RECIST criteria (measured by CT/MRI) | 2.5 years
To evaluate changes in tumor volume (measured by volumetric CT/MRI) | 2.5 years
To evaluate changes in tumor vascularity and to estimate the relationship between dose/pharmacokinetics and vascular response (measured by DCE-MRI) | 2.5 years
To evaluate the incidence of anti-AMG 780 antibody formation | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Los Angeles, California
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio

REFERENCES:
- [Derived] Crockett SD, Barry EL, Mott LA, Snover DC, Wallace K, Baron JA. Predictors of Incident Serrated Polyps: Results from a Large Multicenter Clinical Trial. Cancer Epidemiol Biomarkers Prev. 2022 May 4;31(5):1058-1067. doi: 10.1158/1055-9965.EPI-21-1226. PMID 35506244
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com